CLINICAL TRIAL: NCT04212078
Title: Intracameral Levofloxacin (0.5%) Versus Intracameral Cefuroxime (1mg/0.1ml) Effect on Corneal Endothelial Cell Count and Morphology in Uneventful Phacoemulsification
Brief Title: Intracameral Levofloxacin (0.5%) vs Intracameral Cefuroxime
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National University of Malaysia (Other)
Collaborators: Santen Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Wan Haslina Wan Abdul Halim, Consultant Ophthalmologist-Cornea And Anterior Segment, National University of Malaysia
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: FF-2019-133
Record Dates: First submitted 2019-12-10; First posted 2019-12-26 (Actual); Last update posted 2020-09-21 (Actual); Status verified 2020-09

CONDITIONS: Endophthalmitis Postoperative
Keywords: Intracameral Cefuroxime; Levofloxacin; Corneal Endothelial Cell count; Corneal Morphology
MeSH Terms: interventions — Cefuroxime

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A-Levofloxacin (Active Comparator): 0.1 ml/0.5mg of levofloxacin 0.5% ophthalmic solution
  Interventions: Drug: Levofloxacin Ophthalmic
- B-Intracameral Cefuroxime (Active Comparator): 0.1 ml/1mg of Cefuroxime
  Interventions: Drug: Cefuroxime

INTERVENTIONS:
Drug: Levofloxacin Ophthalmic — 0.1ml which has 0.5 mg levofloxacin will be injected via intracameral into the anterior chamber through the side port wound using a tuberculin syringe in a 27 gauge cannula.
  Other Names: Cravit 0.5%
  Arms: A-Levofloxacin
Drug: Cefuroxime — The vial contains 750 mg of cefuroxime powder is diluted with 7.5 ml of Balanced Salt Solution (BSS). 1 ml of the solution will be withdrawn and added with 9 ml of BSS. Then, 0.1 ml of solution which is equivalent to 1 mg of cefuroxime will be aspirated and kept a side. The dissolution of the antibiotic is confirmed by naked eye. Then the antibiotic of 0.1 ml will be given as intracameral to patient using a tuberculin syringe in a 27 gauge cannula at side port wound at the end of surgery.
  Other Names: Zinacef
  Arms: B-Intracameral Cefuroxime

SUMMARY:
Endophthalmitis is a clinical diagnosis made when intraocular inflammation involving both posterior and anterior chamber; is attributable to bacterial or fungal infection. It is a serious intraocular inflammatory disorder which can be spread via endogenous or exogenous access into the eye by infecting organism. Exogenous spread usually happens post intraocular surgery or procedure (i.e. cataract, vitrectomy, glaucoma filtration surgery) while endogenous spread is associated with hematogenous spread. The occurrence of endophthalmitis accounts for serious post-operative complication which can lead to severe vision loss and even blindness. There are several studies conducted to ascertain the efficiency of intracameral antibiotic as post-operative endophthalmitis prophylaxis. However, there is limited study in human using intracameral levofloxacin to evaluate its effect.This study is designed to compare between intracameral levofloxacin and intracameral cefuroxime in terms of corneal endothelial cell count and its morphology and central corneal thickness in uncomplicated phacoemulsification surgery

DETAILED DESCRIPTION:
This is a prospective, double - blinded randomized clinical trial conducted in University Kebangsaan Malaysia Medical Centre (UKMMC). All patients from Ophthalmology Clinic in UKM Medical Centre from December 2018 till June 2021 will be involved in this study. Patients who fulfill the inclusion criteria will be included in this study.

Preoperative assessment includes proper history taking and ocular examinations.Ocular examination includes baseline visual acuity, slit lamp examinations to ascertain the cataract grading, anterior chamber reactions preoperatively, intraocular pressure measurement via applanation tonometry and fundus examinations using 78D condensing lens. Cornea endothelial examinations will be done by using non-contact TOPCON Specular Microscopy model SP-1P.

On the day of surgery, patients will be informed about the two different antibiotics available that will be used at the end of cataract surgery. A written informed consent will be obtained from the patient.

Patients will be randomized before entering the operating theatre. Sealed envelopes total of 4 will be prepared by the researcher; 2 of which will be labelled as A and another 2 envelopes will be labelled as B. The researcher will randomly pick 1 envelope and allocate to patient's file. The staff nurse in charge will then open the envelope, label A or B will then be pasted on the patient's file (rear part) for documentation.

Cataract surgery will be performed byusing Centurion®Vision System, Alcon, Texas, United Stated of America (USA) phacoemulsification machine. 0.3 ml of levofloxacin 0.5% ophthalmic solution (Cravit®, Santen) will be syringed out and at the conclusion of cataract surgery, the solution of 0.1ml which has 0.5 mg levofloxacin will be injected via intracameral into the anterior chamber through the side port wound using a tuberculin syringe in a 27 gauge cannula.

On the other hand, at the beginning part of surgery, cefuroxime will be diluted by the researcher. In order to reduce dilution error and contamination, dilution will be done strictly according to a standardised protocol that was obtained from Malaysian Clinical Practice Guideline. The vial contains 750 mg of cefuroxime powder is diluted with 7.5 ml of Balanced Salt Solution (BSS). 1 ml of the solution will be withdrawn and added with 9 ml of BSS. Then, 0.1 ml of solution which is equivalent to 1 mg of cefuroxime will be aspirated and kept a side. Then the antibiotic of 0.1 ml will be given as intracameral to patient using a tuberculin syringe in a 27 gauge cannula at side port wound at the end of surgery. The side port wound will then be sealed by stromal hydration and checked for water tightness.

This will be followed by instillation of topical guttae ciprofloxacin 0.3% (Ciloxan, Alcon) and guttae dexamethasone 0.1% (Maxidex, Alcon) and eye shield will be applied before leaving the operating theatre.

Patient will be reviewed again after 2 hours post operatively at the slit lamp and eye drops guttae ciprofloxacin 0.3% and guttae dexamethasone 0.1% will be instilled every 2 hours (5 minutes apart from one eye drop to another) for the first one week post-surgery. Upon discharge, patient will be reviewed again in eye clinic after 1 week and during this visit, these eye drops will then be tapered to 4 hourly for two weeks then six hourly for two weeks until next review. After one month the eye drops will be discontinued.

Patients will then be reviewed after one week, one month and three months post operation. During each visit, patient will be examined under slit lamp to look for anterior chamber reaction and to measure intraocular pressure. They will undergo specular microscopy examination to assess cornea endothelial cell count and morphology and central cornea thickness.

ELIGIBILITY:
Inclusion Criteria:

* All patients with senile cataract and age 50 - 80 years

Exclusion Criteria:

* Patients with cataract other than senile cataract (e.g. traumatic cataract)
* Patients with underlying cornea disease (e.g. cornea dystrophy)
* Patients with corneal endothelial disease/endothelial cell count less than 1000/sqmm².
* Patients with intraoperative complications such as posterior capsule rupture/ prolapsed iris/ zonulysis/ anterior vitreous loss.
* Cataract grading nucleosclerosis (NS) 2+ and below.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Estimated)
Dates: Start 2019-07-29 (Actual); Primary Completion 2022-01 (Estimated); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
Comparison of change in Endothelial cell count concentration in patients treated with intracameral levofloxacin ophthalmic solution and intracameral cefuroxime in an uneventful phacoemulsification. | 1-week post-operation
  Change in Concentration of Endothelial cell count (cells/mm2) from Baseline, measured at 1-week post-operation using a non-contact TOPCON Specular Microscopy model SP-1P.
Comparison of change in Endothelial cell count concentration in patients treated with intracameral levofloxacin ophthalmic solution and intracameral cefuroxime in an uneventful phacoemulsification. | 1-month post-operation
  Change in Concentration of Endothelial cell count (cells/mm2) from Baseline, measured at 1-month post-operation using a non-contact TOPCON Specular Microscopy model SP-1P.
Comparison of change in Endothelial cell count concentration in patients treated with intracameral levofloxacin ophthalmic solution and intracameral cefuroxime in an uneventful phacoemulsification. | 3-month post-operation
  Change in Concentration of Endothelial cell count (cells/mm2) from Baseline, measured at 3-month post-operation using a non-contact TOPCON Specular Microscopy model SP-1P.
Comparison of change in Endothelial cell morphology in patients treated with intracameral levofloxacin ophthalmic solution and intracameral cefuroxime in an uneventful phacoemulsification. | 1-week post-operation
  Change in Endothelial cell morphology from Baseline by assessing the Polymegathism (CV) which is the variation in individual cell areas, and Pleomorphism which is the increased in variability of cell shape, at 1-week post-operation using a non-contact TOPCON Specular Microscopy model SP-1P.
Comparison of change in endothelial cell morphology in patients treated with intracameral levofloxacin ophthalmic solution and intracameral cefuroxime in an uneventful phacoemulsification. | 1-month post-operation
  Change in Endothelial cell morphology from Baseline by assessing the Polymegathism (CV) which is the variation in individual cell areas, and Pleomorphism which is the increased in variability of cell shape, at 1-month post-operation using a non-contact TOPCON Specular Microscopy model SP-1P.
Comparison of change in endothelial cell morphology in patients treated with intracameral levofloxacin ophthalmic solution and intracameral cefuroxime in an uneventful phacoemulsification. | 3-month post-operation
  Change in Endothelial cell morphology from Baseline by assessing the Polymegathism (CV) which is the variation in individual cell areas, and Pleomorphism which is the increased in variability of cell shape, at 3-month post-operation using a non-contact TOPCON Specular Microscopy model SP-1P.
Comparison of change in Central cornea thickness in patients treated with intracameral levofloxacin ophthalmic solution and intracameral cefuroxime in an uneventful phacoemulsification. | 1-week post-operation
  Change in Central cornea thickness (µm) from Baseline, measured at 1-week post-operation using a non-contact TOPCON Specular Microscopy model SP-1P.
Comparison of change in Central cornea thickness in patients treated with intracameral levofloxacin ophthalmic solution and intracameral cefuroxime in an uneventful phacoemulsification. | 1-month post-operation
  Change in Central cornea thickness (µm) from Baseline, measured at 1-month post-operation using a non-contact TOPCON Specular Microscopy model SP-1P.
Comparison of change in Central cornea thickness in patients treated with intracameral levofloxacin ophthalmic solution and intracameral cefuroxime in an uneventful phacoemulsification. | 3-month post-operation
  Change in Central cornea thickness (µm) from Baseline, measured at 3-month post-operation using a non-contact TOPCON Specular Microscopy model SP-1P.
Comparison of Anterior chamber reaction in patients treated with intracameral levofloxacin ophthalmic solution with intracameral cefuroxime in an uneventful phacoemulsification. | 1-week post-operation
  Anterior chamber cell grading refers to presence of inflammatory reaction in the anterior chamber (the space in front of iris plane and cornea endothelium). It is graded by counting the number of cells that is present with slit beam of 1mm x 1mm with high intensity of light measured using the slit lamp at 1-week post-operation.
Comparison of Anterior chamber reaction in patients treated with intracameral levofloxacin ophthalmic solution with intracameral cefuroxime in an uneventful phacoemulsification. | 1-month post-operation
  Anterior chamber cell grading refers to presence of inflammatory reaction in the anterior chamber (the space in front of iris plane and cornea endothelium). It is graded by counting the number of cells that is present with slit beam of 1mm x 1mm with high intensity of light measured using the slit lamp at 1-month post-operation
Comparison of Anterior chamber reaction in patients treated with intracameral levofloxacin ophthalmic solution with intracameral cefuroxime in an uneventful phacoemulsification. | 3-month post-operation
  Anterior chamber cell grading refers to presence of inflammatory reaction in the anterior chamber (the space in front of iris plane and cornea endothelium). It is graded by counting the number of cells that is present with slit beam of 1mm x 1mm with high intensity of light measured using the slit lamp at 3-month post-operation

SECONDARY OUTCOMES:
Side effects | Post-operative period until study completion, an average of 2 years
  To report any untoward incidence of endophthalmitis during the study period.

CONTACTS AND LOCATIONS:
Overall Officials: Wan Haslina Wan Abdul Halim, M.D, Study Chair — Department of Ophthalmology, UKM Medical Centre
Locations (1):
- UKM Medical Centre, Kuala Lumpur, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kernt M, Kampik A. Endophthalmitis: Pathogenesis, clinical presentation, management, and perspectives. Clin Ophthalmol. 2010 Mar 24;4:121-35. doi: 10.2147/opth.s6461. PMID 20390032
- [Background] Lee MY, Goh PP, Salowi MA, Adnan TH, Ismail M. The Malaysian Cataract Surgery Registry: Cataract Surgery Practice Pattern. Asia Pac J Ophthalmol (Phila). 2014 Nov-Dec;3(6):343-7. doi: 10.1097/APO.0000000000000030. PMID 26107976
- [Background] Lockington D, Flowers H, Young D, Yorston D. Assessing the accuracy of intracameral antibiotic preparation for use in cataract surgery. J Cataract Refract Surg. 2010 Feb;36(2):286-9. doi: 10.1016/j.jcrs.2009.08.034. PMID 20152612
- [Background] Espiritu CR, Caparas VL, Bolinao JG. Safety of prophylactic intracameral moxifloxacin 0.5% ophthalmic solution in cataract surgery patients. J Cataract Refract Surg. 2007 Jan;33(1):63-8. doi: 10.1016/j.jcrs.2006.09.019. PMID 17189795
- [Background] Endophthalmitis Study Group, European Society of Cataract & Refractive Surgeons. Prophylaxis of postoperative endophthalmitis following cataract surgery: results of the ESCRS multicenter study and identification of risk factors. J Cataract Refract Surg. 2007 Jun;33(6):978-88. doi: 10.1016/j.jcrs.2007.02.032. PMID 17531690
- [Background] Montan PG, Wejde G, Setterquist H, Rylander M, Zetterstrom C. Prophylactic intracameral cefuroxime. Evaluation of safety and kinetics in cataract surgery. J Cataract Refract Surg. 2002 Jun;28(6):982-7. doi: 10.1016/s0886-3350(01)01270-6. PMID 12036640
- [Background] Friling E, Lundstrom M, Stenevi U, Montan P. Six-year incidence of endophthalmitis after cataract surgery: Swedish national study. J Cataract Refract Surg. 2013 Jan;39(1):15-21. doi: 10.1016/j.jcrs.2012.10.037. PMID 23245359
- [Background] Raen M, Sandvik GF, Drolsum L. Endophthalmitis following cataract surgery: the role of prophylactic postoperative chloramphenicol eye drops. Acta Ophthalmol. 2013 Mar;91(2):118-22. doi: 10.1111/j.1755-3768.2011.02324.x. Epub 2011 Dec 13. PMID 22151787
- [Background] Shahraki K, Fard MNA, Shahri F, Pourmatin R, Mohammadi T, Boroumand PG, Shahraki K. Effects of intracameral cefuroxime on corneal endothelial cell counts and its morphology after cataract surgery. Interv Med Appl Sci. 2017 Jun;9(2):100-104. doi: 10.1556/1646.9.2017.2.13. PMID 28932504
- [Background] Cakir B, Celik E, Aksoy NO, Bursali O, Ucak T, Bozkurt E, Alagoz G. Toxic anterior segment syndrome after uncomplicated cataract surgery possibly associated with intracamaral use of cefuroxime. Clin Ophthalmol. 2015 Mar 17;9:493-7. doi: 10.2147/OPTH.S74249. eCollection 2015. PMID 25834384
- [Background] Louis B.Cantor, Christopher J. Rapuano, George A. Cioffi. Basic and Clinical Science Course. Section 9: Intraocular inflammation and uveitis. American Academy of Ophthalmology 2014-2015;8;261.
- [Background] Management of Post-operative Infectious Endophthalmitis. Clinical Practice Guideline. August 2006. Ministry of Health Malaysia.
- [Background] Matsuura K, Miyoshi T, Suto C, Akura J, Inoue Y. Efficacy and safety of prophylactic intracameral moxifloxacin injection in Japan. J Cataract Refract Surg. 2013 Nov;39(11):1702-6. doi: 10.1016/j.jcrs.2013.05.036. Epub 2013 Sep 18. PMID 24054967
- [Background] Mather R, Karenchak LM, Romanowski EG, Kowalski RP. Fourth generation fluoroquinolones: new weapons in the arsenal of ophthalmic antibiotics. Am J Ophthalmol. 2002 Apr;133(4):463-6. doi: 10.1016/s0002-9394(02)01334-x. PMID 11931779
- [Background] Kim SY, Park YH, Lee YC. Comparison of the effect of intracameral moxifloxacin, levofloxacin and cefazolin on rabbit corneal endothelial cells. Clin Exp Ophthalmol. 2008 May;36(4):367-70. doi: 10.1111/j.1442-9071.2008.01771.x. PMID 18700925
- [Background] Kanda Y, Kayama T, Okamoto S, et al. A post-marketing surveillance of 0.5% levofloxacin ophthalmic solution for external ocular infections [in Japanese]. Rinsho Ganka 2008; 62 (13): 2007-17.
- [Background] Pea F, Ferrari E, Pavan F, Roman-Pognuz D, Bandello F, Furlanut M. Levofloxacin disposition over time in aqueous humor of patients undergoing cataract surgery. Antimicrob Agents Chemother. 2005 Jun;49(6):2554-7. doi: 10.1128/AAC.49.6.2554-2557.2005. PMID 15917572
- [Background] Keating GM. Levofloxacin 0.5% ophthalmic solution: a review of its use in the treatment of external ocular infections and in intraocular surgery. Drugs. 2009 Jun 18;69(9):1267-86. doi: 10.2165/00003495-200969090-00009. PMID 19537841
- [Background] Matsuura K, Mori T, Miyamoto T, Suto C, Saeki Y, Tanaka S, Kawamura H, Ohkubo S, Tanito M, Inoue Y. Survey of Japanese ophthalmic surgeons regarding perioperative disinfection and antibiotic prophylaxis in cataract surgery. Clin Ophthalmol. 2014 Sep 29;8:2013-8. doi: 10.2147/OPTH.S64756. eCollection 2014. PMID 25302013
- [Background] Choi JA, Chung SK. Safety of intracameral injection of gatifloxacin, levofloxacin on corneal endothelial structure and viability. J Ocul Pharmacol Ther. 2009 Oct;25(5):425-31. doi: 10.1089/jop.2009.0010. PMID 19857104
- [Background] Espiritu CRG, Bolinao JG. Prophylactic intracameral levofloxacin in cataract surgery - an evaluation of safety. Clin Ophthalmol. 2017 Dec 12;11:2199-2204. doi: 10.2147/OPTH.S144625. eCollection 2017. PMID 29276375
- [Background] Louis B.Cantor, Christopher J. Rapuano, George A. Cioffi. Basic and Clinical Science Course. Section 8: External Disease and Cornea. American Academy of Opthalmology 2016-2017; 1; 6-9.
- [Background] Louis B.Cantor, Christopher J. Rapuano, George A. Cioffi. Basic and Clinical Science Course. Section 11: Lens and Cataract. American Academy of Ophthalmology 2014-2015; 8; 146-151.
- [Background] Duman R, Tok Cevik M, Gorkem Cevik S, Duman R, Perente I. Corneal endothelial cell density in healthy Caucasian population. Saudi J Ophthalmol. 2016 Oct-Dec;30(4):236-239. doi: 10.1016/j.sjopt.2016.10.003. Epub 2016 Nov 2. PMID 28003782
- [Background] Ganekal S, Nagarajappa A. Comparison of morphological and functional endothelial cell changes after cataract surgery: phacoemulsification versus manual small-incision cataract surgery. Middle East Afr J Ophthalmol. 2014 Jan-Mar;21(1):56-60. doi: 10.4103/0974-9233.124098. PMID 24669147
- [Background] Reuschel A, Bogatsch H, Barth T, Wiedemann R. Comparison of endothelial changes and power settings between torsional and longitudinal phacoemulsification. J Cataract Refract Surg. 2010 Nov;36(11):1855-61. doi: 10.1016/j.jcrs.2010.06.060. PMID 21029892
- [Background] Liu Y, Zeng M, Liu X, Luo L, Yuan Z, Xia Y, Zeng Y. Torsional mode versus conventional ultrasound mode phacoemulsification: randomized comparative clinical study. J Cataract Refract Surg. 2007 Feb;33(2):287-92. doi: 10.1016/j.jcrs.2006.10.044. PMID 17276271
- [Background] Walkow T, Anders N, Klebe S. Endothelial cell loss after phacoemulsification: relation to preoperative and intraoperative parameters. J Cataract Refract Surg. 2000 May;26(5):727-32. doi: 10.1016/s0886-3350(99)00462-9. PMID 10831904
- [Background] Storr-Paulsen A, Norregaard JC, Farik G, Tarnhoj J. The influence of viscoelastic substances on the corneal endothelial cell population during cataract surgery: a prospective study of cohesive and dispersive viscoelastics. Acta Ophthalmol Scand. 2007 Mar;85(2):183-7. doi: 10.1111/j.1600-0420.2006.00784.x. PMID 17305732
- [Background] Hayashi K, Hayashi H, Nakao F, Hayashi F. Risk factors for corneal endothelial injury during phacoemulsification. J Cataract Refract Surg. 1996 Oct;22(8):1079-84. doi: 10.1016/s0886-3350(96)80121-0. PMID 8915805
- [Background] Chang A, Fridberg A, Kugelberg M. Comparison of phacoemulsification cataract surgery with low versus standard fluidic settings and the impact on postoperative parameters. Eur J Ophthalmol. 2017 Jan 19;27(1):39-44. doi: 10.5301/ejo.5000813. Epub 2016 May 31. PMID 27312207
- [Background] Hasegawa Y, Nejima R, Mori Y, Sakisaka T, Minami K, Miyata K, Oshika T. Risk factors for corneal endothelial cell loss by cataract surgery in eyes with pseudoexfoliation syndrome. Clin Ophthalmol. 2016 Aug 30;10:1685-9. doi: 10.2147/OPTH.S106661. eCollection 2016. PMID 27621588
- [Background] Doerte Luensmann. The Endothelium - What Difference do SiH Lenses Make? High-Dk silicone Hydrogel lenses. May 2010.
- [Background] Chylack LT Jr, Wolfe JK, Singer DM, Leske MC, Bullimore MA, Bailey IL, Friend J, McCarthy D, Wu SY. The Lens Opacities Classification System III. The Longitudinal Study of Cataract Study Group. Arch Ophthalmol. 1993 Jun;111(6):831-6. doi: 10.1001/archopht.1993.01090060119035. PMID 8512486
- [Background] The Standardisation of Uveitis Nomenclature (SUN) Working Group. Grading Scheme for Anterior Chamber Cells.
- [Background] Julious SA. Sample sizes for clinical trials with normal data. Stat Med. 2004 Jun 30;23(12):1921-86. doi: 10.1002/sim.1783. PMID 15195324